CLINICAL TRIAL: NCT05987670
Title: Triple Cardiovascular Disease Detection With an Artificial Intelligence-enabled Stethoscope
Acronym: TRICORDER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Health Partners (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22HH8045
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Heart Valve Diseases; Atrial Fibrillation; Heart Murmurs; Congestive Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: cluster randomized controlled trial; artificial intelligence; digital health; cardiology; primary care
MeSH Terms: conditions — Heart Failure; Heart Valve Diseases; Atrial Fibrillation; Heart Murmurs

STUDY DESIGN:
Intervention Model Description: Open label cluster randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Receive 3-6 AI-stethoscopes (Eko DUO, Eko Health Inc, CA, USA) including artificial intelligence software for detection of:
  1. Reduced left ventricular ejection fraction <40%
  2. Atrial fibrillation
  3. Cardiac murmurs
  Interventions: Device: AI-stethoscope
- Control (No Intervention): Usual care

INTERVENTIONS:
Device: AI-stethoscope — Clinicians at practices in the intervention arm will be provided with one session of in-person training in use of the AI-stethoscope within 2 weeks of randomisation, including
  1. Delivery and setup
  2. Smartphone app installation and login
  3. Pairing of all clinician smartphones with all AI-stethoscopes in the same practice
  4. Demo of patient examination The AI-stethoscope will be used within its CE/UKCA-marked intended purpose. The clinical guidelines for use have been agreed by the NHS North West London Integrated Care System and Betsi Cadwaladr University Health Board Cardiovascular Executive Groups. Patients will be examined with the AI-stethoscope in accordance with these guidelines, and/or where stethoscope examination is deemed clinically appropriate. Patients will provide verbal consent for examination with the AI-stethoscope as per any physical examination performed by healthcare professionals for direct care, in accordance with UK law and General Medical Council guidelines.
  Other Names: Eko DUO; Eko Core 500; Eko EAS
  Arms: Intervention

SUMMARY:
Heart failure (HF) is a condition in which the heart cannot pump blood adequately. It is increasingly common, consumes 4% of the UK National Health Service (NHS) budget and is deadlier than most cancers. Early diagnosis and treatment of HF improves quality of life and survival. Unacceptably, 80% of patients have their HF diagnosed only when very unwell, requiring an emergency hospital admission, with worse survival and higher treatment costs to the NHS. This is largely because General Practitioners (GPs) have no easy-to-use tools to check for suspected HF, with patients having to rely on a long and rarely completed diagnostic pathway involving blood tests and hospital assessment.

The investigators have previously demonstrated that an artificial intelligence-enabled stethoscope (AI-stethoscope) can detect HF in 15 seconds with 92% accuracy (regardless of age, gender or ethnicity) - even before patients develop symptoms. While the GP uses the stethoscope, it records the heart sounds and electrical activity, and uses inbuilt artificial intelligence to detect HF.

The goal of this clinical trial is to determine the clinical and cost-effectiveness of providing primary care teams with the AI-stethoscope for the detection of heart failure. The main questions it aims to answer are if provision of the AI-stethoscope:

1. Increases overall detection of heart failure
2. Reduces the proportion of patients being diagnosed with heart failure following an emergency hospital admission
3. Reduces healthcare system costs

200 primary care practices across North West London and North Wales, UK, will be recruited to a cluster randomised controlled trial, meaning half of the primary care practices will be randomly assigned to have AI-stethoscopes for use in direct clinical care, and half will not. Researchers will compare clinical and cost outcomes between the groups.

DETAILED DESCRIPTION:
Triple Cardiovascular Disease Detection with Artificial Intelligence-enabled Stethoscope (TRICORDER) is an open label, cluster randomised controlled trial. The aim is to determine whether use of an artificial intelligence-enabled stethoscope (AI-stethoscope) in UK Primary Care improves community-based detection of heart failure (HF), compared with usual care. 200 primary care practices in North West London (UK) will be randomised to receive the AI-stethoscope (intervention arm) or continue with usual care (control arm). The intervention arm will use the AI-stethoscope in routine clinical practice. Outcomes will be measured using pooled primary and secondary care clinical and cost-data, as well as clinician questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practices that care for adult patients and have the ability to request natriuretic peptide blood testing
* Primary care practices within the NIHR North West London Clinical Research Network or Betsi Cadwaladr University Health Board.

Exclusion Criteria:

* Poor WiFi and/or mobile data connectivity within primary care consulting rooms
* No face-to-face patient consultations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of heart failure (co-primary) | 24 months
  Difference in incidence of coded new diagnoses of heart failure (HF)
Ratio of route to diagnosis of heart failure (co-primary) between emergency and community-based pathways | 24 months
  Difference in ratio of the incidence of coded diagnoses of HF via hospital admission-based versus community-based pathways.

SECONDARY OUTCOMES:
Incidence of atrial fibrillation | 24 months
  New coded diagnoses of atrial fibrillation (AF)
Incidence of valvular heart disease | 24 months
  New coded diagnoses of valvular heart disease (VHD)
Cost-consequence (AF) | 24 months
  Cost-consequence analysis (form of health economic evaluation) for diagnosis of atrial fibrillation, stratified by route to diagnosis. Presented in pounds sterling.
Cost-consequence (HFrEF) | 24 months
  Cost-consequence analysis (form of health economic evaluation) for diagnosis of HFrEF, stratified by route to diagnosis. Presented in pounds sterling.
Cost-consequence (VHD) | 24 months
  Cost-consequence analysis (form of health economic evaluation) for diagnosis of VHD, stratified by route to diagnosis. Presented in pounds sterling.
Health service utilisation | 24 months
  Health service utilisation for diagnostics e.g. rates of request for echocardiography, electrocardiography, primary care appointments. Collected from NHS organisation business intelligence repositories and UK Trusted Research Environments.
Proportion of patients prescribed guideline-directed medical therapy | 24 months
  Proportion of patients prescribedguideline-directed medical therapy (HF, AF, VHD)
Device therapy | 24 months
  New implantation of cardiac resynchronisation therapy (CRT) and/or implantable cardioverter-defibrillator (ICD)
Uptake and utilisation | 24 months
  Differential rates of uptake and utilisation of AI-stethoscope in primary care
Determinants of uptake and utilisation | 24 months
  Determinants of utilisation of AI-stethoscope in primary care (clinician questionnaires)
Patient quality of life | 24 months
  Healthy Days at Home (patient-level analysis)

OTHER OUTCOMES:
Sensitivity analysis | 24 months
  Patient-level sensitivity analyses will be performed for patients with abnormal Eko DUO predictions for HF, to identify direct associations between AI-stethoscope predictions and specific diagnostic codes for HF, AF and VHD

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Peters, MD, Principal Investigator — Imperial College London
Locations (1):
- NHS North West London Integrated Care System, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bachtiger P, Petri CF, Scott FE, Ri Park S, Kelshiker MA, Sahemey HK, Dumea B, Alquero R, Padam PS, Hatrick IR, Ali A, Ribeiro M, Cheung WS, Bual N, Rana B, Shun-Shin M, Kramer DB, Fragoyannis A, Keene D, Plymen CM, Peters NS. Point-of-care screening for heart failure with reduced ejection fraction using artificial intelligence during ECG-enabled stethoscope examination in London, UK: a prospective, observational, multicentre study. Lancet Digit Health. 2022 Feb;4(2):e117-e125. doi: 10.1016/S2589-7500(21)00256-9. Epub 2022 Jan 5. PMID 34998740
- [Background] Bachtiger P, Kelshiker MA, Petri CF, Gandhi M, Shah M, Kamalati T, Khan SA, Hooper G, Stephens J, Alrumayh A, Barton C, Kramer DB, Plymen CM, Peters NS. Survival and health economic outcomes in heart failure diagnosed at hospital admission versus community settings: a propensity-matched analysis. BMJ Health Care Inform. 2023 Mar;30(1):e100718. doi: 10.1136/bmjhci-2022-100718. PMID 36921978
- [Derived] Kelshiker MA, Bachtiger P, Mansell J, Kramer DB, Nakhare S, Almonte MT, Alrumayh A, Petri CF, Peters A, Costelloe C, Falaschetti E, Barton C, Al-Lamee R, Majeed A, Plymen CM, Peters NS. Triple cardiovascular disease detection with an artificial intelligence-enabled stethoscope (TRICORDER): design and rationale for a decentralised, real-world cluster-randomised controlled trial and implementation study. BMJ Open. 2025 May 21;15(5):e098030. doi: 10.1136/bmjopen-2024-098030. PMID 40398956